CLINICAL TRIAL: NCT02972996
Title: Effects of Blueberry Consumption on Cardiometabolic Parameters in Men With Type 2 Diabetes.
Brief Title: Blueberry Consumption and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HNS 01
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Results first posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-02

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — blueberry extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blueberry (Experimental): 22 g freeze-dried blueberries
  Interventions: Other: Blueberry
- Placebo (Placebo Comparator): 22 g placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Blueberry — 22 g freeze-dried whole blueberry powder
  Arms: Blueberry
Other: Placebo — 22 g placebo blueberry powder
  Arms: Placebo

SUMMARY:
Lifestyle strategies that include dietary modification, such as consumption of a plant-based diet, are well recognized in disease prevention and may improve type 2 diabetes. Various components of a plant-based diet may contribute to its beneficial health effects, but there has been keen interest in the possibility that plant polyphenols may have a role. Blueberries are dietary sources of polyphenols, specifically anthocyanins. To date there are few human clinical trials evaluating the beneficial health effects of blueberries in populations with type 2 diabetes. The objective of the study is to determine if freeze-dried blueberries compared to a blueberry placebo will improve cardiometabolic parameters in men with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Ages 45 to 75 years at beginning of study
* BMI >25 kg/m2
* HbA1C > 6.5 and < 9
* Medical diagnosis of type 2 diabetes for at least 6 months

Exclusion Criteria:

* Use of insulin
* Presence of chronic kidney disease (GFR < 45 mL/min), liver cirrhosis, gastrointestinal disease, pancreatic disease, or malabsorption syndromes
* Weight loss of >10% of body weight over the last 6 months; routine participation in heavy exercise
* Heavy smokers (>20 cigarettes per day)
* Unable or unwilling to give informed consent or communicate with study staff
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigators may interfere with study participation or the ability to follow the intervention protocol
* Allergies to blueberries or blueberry products

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret M. Wilson, MS, RD, CDE, Principal Investigator — Stratton V.A. Medical Center
Locations (1):
- Stratton V.A. Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stote KS, Wilson MM, Hallenbeck D, Thomas K, Rourke JM, Sweeney MI, Gottschall-Pass KT, Gosmanov AR. Effect of Blueberry Consumption on Cardiometabolic Health Parameters in Men with Type 2 Diabetes: An 8-Week, Double-Blind, Randomized, Placebo-Controlled Trial. Curr Dev Nutr. 2020 Mar 9;4(4):nzaa030. doi: 10.1093/cdn/nzaa030. eCollection 2020 Apr. PMID 32337475

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blueberry | Placebo
Started | 27 | 28
Completed | 26 | 26
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blueberry | Placebo | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (1.1) | 66.7 (1.1) | 67.0 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 26 | 26 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 25 | 24 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Blood Pressure [Mean (Standard Deviation); unit: mm Hg]
  Systolic blood pressure | 130.3 (21.7) | 126.2 (13.3) | 128.2 (18.0)
  Diastolic blood pressure | 73.4 (5.4) | 76.2 (7.8) | 74.8 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure
Description: Systolic blood pressure and diastolic blood pressure.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Blueberry | Placebo
Number analyzed (Participants) | 26 | 26
mm Hg
  Systolic blood pressure | 125.6 (2.5) | 126.0 (2.5)
  Diastolic blood pressure | 74.6 (1.0) | 75.1 (1.0)
Statistical Analysis 1: Comparison: Blueberry vs Placebo; Values are least-squares means ± SEs (adjusted for the baseline values) from ANCOVA linear mixed model that included covariates of age, baseline (pretreatment values), BMI and weight; Test type: Other; p = 0.56, ANCOVA

2. Secondary Outcome: Hemoglobin A1C
Description: Hemoglobin A1C is a surrogate marker of glycemic control over the preceding 2-3 months.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Blueberry | Placebo
Number analyzed (Participants) | 26 | 26
percent | 7.1 (0.1) | 7.5 (0.2)
Statistical Analysis 1: Comparison: Blueberry vs Placebo; Test type: Other; p = 0.03, ANCOVA

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Blueberry | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT02972996/Prot_SAP_000.pdf